CLINICAL TRIAL: NCT00473733
Title: Glucagon Like Peptides Receptors Expression in the Stomach of Diabetes Type 2
Acronym: GLP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 65/07
Record Dates: First submitted 2007-05-13; First posted 2007-05-15 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus Type 2
Keywords: PATIENTS WITH DIABETES MELLITUS TYPE 2; UNDERGO UPPER ENDOSCOPY; BIOPSIES FOR GLP RECEPTORS EXPRESSION; PCR ANALYSIS
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Endoscopy, Digestive System

INTERVENTIONS:
Procedure: GLP receptors expression
Procedure: ESOPHAGOGASTRODUODENOSCOPY

SUMMARY:
Glucagon like peptides receptors expression in the stomach of diabetes type 2 Glucagon like peptides (GLP-1, GLP-2), are hormones secreted by L cells located along the gastrointestinal tract. These hormones are secreted after meals and have some roles in regulating the digestion process, absorption, and sending signals to the brain that regulate food consumption. GLP peptides affect peripheral targets and have an important homeostatic role. GLP-1 decreases the circulatory glucose level and GLP-2 has trophic effects which enable adequate intestine growth.

We aimed in our study to investigate the GLP-1 and GLP-2 receptor expression in different zones of the stomach in diabetes type 2 patients. If there are differences, it might explain the pathological gastric emptying in these patients.

Understanding the function of these peptides may lead to new therapeutic options for diabetic patients with delayed gastric emptying.

Methods: 20 diabetes type 2 patients with symptoms that need upper endoscopy will be included in the study and 20 controls aged 18-70 years. Patients with neurological disease will be excluded. During esophagogastroduodenoscopy 3 biopsies will be taken from the antrum, corpus and cardia. The biopsies will be stored in -70. After RNA extraction the GLP receptors expression will established by real time PCR method. Patients with different expression compared to control will undergo isotopic scan for gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* 20 diabetes type 2 patients with symptoms that need upper endoscopy will be included in the study and 20 controls aged 18-70 years

Exclusion Criteria:

* Patients with neurological disease will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Broide, MD, Principal Investigator — Ethic committee of Asaaf Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel